CLINICAL TRIAL: NCT03837574
Title: French National Registry of Patients With Tetralogy of Fallot and Implantable Cardioverter Defibrillator
Acronym: DAI-T4F
Status: Recruiting | Type: Observational
Sponsor: Paris Sudden Death Expertise Center (Other)
Responsible Party: Principal Investigator, Marijon, Principal Investigator Dr Victor WALDMANN, Paris Sudden Death Expertise Center
Other Study IDs: CNIL2029070
Record Dates: First submitted 2019-01-27; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Tetralogy of Fallot; Implantable Defibrillator User; Congenital Heart Disease; Sudden Cardiac Death; Ventricular Arrythmia
Keywords: tretalogy of fallot; implantable cardioverter defibrillator; congenital heart disease; sudden cardiac death; ventricular arrhythmia
MeSH Terms: conditions — Tetralogy of Fallot; Heart Defects, Congenital; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
National french registry of patients with tetralogy of Fallot and implantable cardioverter defibrillator.

DETAILED DESCRIPTION:
Inclusion criteria:

* patient with tetralogy of Fallot > 18 years
* implantable cardioverter defibrillator (ICD)
* primary or secondary prevention

All french centers performing ICD implantation are annually contacted to include all patients with tetralogy of Fallot and ICD.

Retrospective inclusion of cases before 2010 and prospective inclusion after 2010 with prospective follow up and annual update.

All events are centrally adjudicated with collection of all baseline ECG and reviewing of endocavitary EGM.

ELIGIBILITY:
Inclusion Criteria:

* tetralogy of Fallot
* implantable cardioverter defibrillator

Exclusion Criteria:

* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with tetralogy of Fallot and implantablle cardioverter defibrillator in France
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-12-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Ventricular arrhythmias | through study completion, an average of 1 year
  Rate of appropriate ICD therapies for ventricular tachycardia and fast ventricular tachycardia / ventricular fibrillation
Complications of ICD | through study completion, an average of 1 year
  Rate of complications of ICD including inappropriate therapies, infection, lead or generator dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Victor Waldmann, MD, Principal Investigator — Paris Sudden Death Expertise Center
Locations (1):
- Paris Sudden Death Expertise Center, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laredo M, Duthoit G, Sacher F, Anselme F, Audinet C, Bessiere F, Bordachar P, Bouzeman A, Boveda S, Bun SS, Chassignolle M, Clerici G, Da Costa A, de Guillebon M, Defaye P, Elbaz N, Eschalier R, Extramiana F, Fauchier L, Hermida A, Gandjbakhch E, Garcia R, Gourraud JB, Guenancia C, Guy-Moyat B, Irles D, Iserin L, Jourda F, Koutbi L, Labombarda F, Ladouceur M, Lagrange P, Lellouche N, Mansourati J, Marquie C, Martins R, Massoulie G, Mathiron A, Maury P, Messali A, Milhem A, Mondoly P, Nguyen C, Ninni S, Pasquie JL, Pierre B, Pujadas P, Sellal JM, Thambo JB, Walton C, Winum P, Zakine C, Zhao A, Jouven X, Combes N, Marijon E, Waldmann V; DAI-T4F Investigators. Rapid ventricular tachycardia in patients with tetralogy of Fallot and implantable cardioverter-defibrillator: Insights from the DAI-T4F nationwide registry. Heart Rhythm. 2023 Feb;20(2):252-260. doi: 10.1016/j.hrthm.2022.10.016. Epub 2022 Oct 26. PMID 36309156
- [Derived] Waldmann V, Bouzeman A, Duthoit G, Koutbi L, Bessiere F, Labombarda F, Marquie C, Gourraud JB, Mondoly P, Sellal JM, Bordachar P, Hermida A, Al Arnaout A, Anselme F, Audinet C, Bernard Y, Boveda S, Bun SS, Chassignolle M, Clerici G, Da Costa A, de Guillebon M, Defaye P, Elbaz N, Eschalier R, Garcia R, Guenancia C, Guy-Moyat B, Halimi F, Irles D, Iserin L, Jourda F, Ladouceur M, Lagrange P, Laredo M, Mansourati J, Massoulie G, Mathiron A, Maury P, Messali A, Narayanan K, Nguyen C, Ninni S, Perier MC, Pierre B, Pujadas P, Sacher F, Sagnol P, Sharifzadehgan A, Walton C, Winum P, Zakine C, Fauchier L, Martins R, Pasquie JL, Thambo JB, Jouven X, Combes N, Marijon E. Sex Differences in Outcomes of Tetralogy of Fallot Patients With Implantable Cardioverter-Defibrillators. JACC Clin Electrophysiol. 2022 Oct;8(10):1304-1314. doi: 10.1016/j.jacep.2022.06.024. Epub 2022 Sep 28. PMID 36266008
- [Derived] Waldmann V, Marquie C, Bouzeman A, Duthoit G, Thambo JB, Koutbi L, Maltret A, Pasquie JL, Combes N, Marijon E. Subcutaneous vs Transvenous Implantable Cardioverter-Defibrillator Therapy in Patients With Tetralogy of Fallot. J Am Coll Cardiol. 2022 Oct 25;80(17):1701-1703. doi: 10.1016/j.jacc.2022.08.761. No abstract available. PMID 36265962
- [Derived] Bessiere F, Gardey K, Bouzeman A, Duthoit G, Koutbi L, Labombarda F, Marquie C, Gourraud JB, Mondoly P, Sellal JM, Bordachar P, Hermida A, Anselme F, Asselin A, Audinet C, Bernard Y, Boveda S, Chevalier P, Clerici G, da Costa A, de Guillebon M, Defaye P, Eschalier R, Garcia R, Guenancia C, Guy-Moyat B, Henaine R, Irles D, Iserin L, Jourda F, Ladouceur M, Lagrange P, Laredo M, Mansourati J, Massoulie G, Mathiron A, Maury P, Nguyen C, Ninni S, Perier MC, Pierre B, Sacher F, Walton C, Winum P, Martins R, Pasquie JL, Thambo JB, Jouven X, Combes N, Di Filippo S, Marijon E, Waldmann V. Impact of Pulmonary Valve Replacement on Ventricular Arrhythmias in Patients With Tetralogy of Fallot and Implantable Cardioverter-Defibrillator. JACC Clin Electrophysiol. 2021 Oct;7(10):1285-1293. doi: 10.1016/j.jacep.2021.02.022. Epub 2021 Apr 28. PMID 33933408
- [Derived] Waldmann V, Bouzeman A, Duthoit G, Koutbi L, Bessiere F, Labombarda F, Marquie C, Gourraud JB, Mondoly P, Sellal JM, Bordachar P, Hermida A, Anselme F, Asselin A, Audinet C, Bernard Y, Boveda S, Bru P, Bun SS, Clerici G, Da Costa A, de Guillebon M, Defaye P, Elbaz N, Eschalier R, Garcia R, Guenancia C, Guy-Moyat B, Halimi F, Irles D, Iserin L, Jourda F, Ladouceur M, Lagrange P, Laredo M, Mansourati J, Massoulie G, Mathiron A, Maury P, Messali A, Narayanan K, Nguyen C, Ninni S, Perier MC, Pierre B, Pujadas P, Sacher F, Sagnol P, Sharifzadehgan A, Walton C, Winum P, Zakine C, Fauchier L, Martins R, Pasquie JL, Thambo JB, Jouven X, Combes N, Marijon E; DAI-T4F Investigators*. Long-Term Follow-Up of Patients With Tetralogy of Fallot and Implantable Cardioverter Defibrillator: The DAI-T4F Nationwide Registry. Circulation. 2020 Oct 27;142(17):1612-1622. doi: 10.1161/CIRCULATIONAHA.120.046745. Epub 2020 Oct 1. PMID 32998542